CLINICAL TRIAL: NCT06526156
Title: The Anesthetic and Recovery Profiles of Low-dose Hypobaric Bupivacaine in Spinal Anesthesia Injected in the L5-S1 Space for Total Hip and Knee Arthroplasty
Brief Title: Hypobaric L5-S1 Study
Status: Active, not recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 24-5192; CAPCR# 24-5192 (Other: UHN)
Record Dates: First submitted 2024-07-11; First posted 2024-07-29 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Anesthesia; Anesthesia, Local
Keywords: Total Hip Arthroplasty; Total Knee Arthroplasty; Bupivacaine
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hypobaric L5-S1 Spinal Anesthesia: Will receive a dose of hypobaric (0.33%) bupivacaine, administered at the L5-S1 space.
  Interventions: Drug: Bupivacaine injection

INTERVENTIONS:
Drug: Bupivacaine injection — A 3 mL hypobaric (0.33%) solution of bupivacaine, prepared by mixing 2 mL of isobaric (0.5%) bupivacaine with 1 mL of sterile water. Dural puncture will be performed using a 25 or 27G (gauge) spinal needle at the L5-S1 intervertebral space, and the 3 mL of 0.33% bupivacaine will be injected into the intrathecal space.
  Other Names: Marcaine

SUMMARY:
Patients going through total hip or knee replacement (arthroplasty) have to be put under spinal anesthesia to prevent them from feeling any pain during surgery. Spinal anesthesia means having a small needle inserted between the bones of the lower lumbar spine (vertebrae). The choice of space used is decided by the anesthesiologist in charge of patient care. The space between these bones is often narrowed by arthritis or other age-related degenerative spine disease in patients having total hip or knee replacement surgery. The lowest L5-S1 (Lumbar 5- Sacral 1) space is the largest one and often least affected by arthritis, which makes it the easiest option. Despite this, it is not currently the most common space used for spinal anesthesia, because it is hard to find by palpation (feeling the bones through the skin), and because there is concern that local anesthetic will not always spread up high enough from this lowest space, which is needed for a successful spinal anesthesia. How far it spreads depends on the amount (dose) and density of local anesthetic given.

There are two types of local anesthetic: one called isobaric, which has the same density as CSF (Cerebro-Spinal Fluid), and another called hypobaric, which has lower density than CSF.

Isobaric local anesthetic spreads evenly throughout the CSF irrespective of patient positioning. However, a larger dose is required to achieve adequate anesthesia for surgery. Using larger doses, leads to a very long duration of sensory and motor block, far in excess of that required for surgical completion which leads to a slower recovery from anesthesia.

Hypobaric local anesthetic, on the other hand, floats in CSF like oil on water. This allows anesthesiologists to use a smaller dose while still being sure that it will spread high enough to achieve adequate anesthesia for surgery. The smaller doses in turn allow for faster recovery of normal movement and feeling in the legs of patients after surgery.

It has been observed that all of these dilemma can be solved by:

1. Using ultrasound imaging to find and mark the space, and
2. Injecting hypobaric local anesthetic.

The goal of this observational study is to determine the success rate of spinal anesthesia with a lower dose of hypobaric bupivacaine injected into the L5-S1 space, when done on total hip or knee arthroplasty patients at Toronto Western Hospital.

DETAILED DESCRIPTION:
Spinal anesthesia is the recommended type of anesthesia for total hip or knee arthroplasty, as it is associated with superior clinical outcomes compared to general anesthesia. However, many patients undergoing these surgical procedures have age-related spine disease, previous spine surgery, or other spinal deformities which make the injection of spinal anesthesia difficult.

One strategy is to administer the spinal anesthesia at the L5-S1 space: it is least affected by arthritic and degenerative changes, and as it is the largest intervertebral space, it has the lowest chance of causing spinal cord trauma.

However, administration of spinal anesthesia at the lowest lumbar intervertebral levels significantly decreases the odds of success of surgical anesthesia. This is due to the fact that the standard solution of 0.5% bupivacaine is isobaric with respect to the cerebrospinal fluid (CSF), leading to unpredictable distribution within the CSF and inconsistent extent of sensory block. It has been shown that an inordinately large dose of 25 mg (5 milliliter) of 0.5% bupivacaine is required to achieve the adequate extent of sensory loss, as opposed to more conventional doses of 12-15 mg (milligram). However, this leads to a very long duration of sensory and motor block, far in excess of that required for surgical completion. This delays patient discharge from the post-anesthetic recovery unit, mobilization, and recovery. This is at odds with the goals of modern total hip and knee arthroplasty, which emphasizes same-day mobilization, physiotherapy, and even same-day hospital discharge. Using lower doses of isobaric bupivacaine, on the other hand, increases the risk of inadequate or failed spinal anesthesia, requiring conversion to general anesthesia.

One strategy to address this dilemma, which has been employed with great success to date at the Toronto Western Hospital (TWH), is to use a solution of bupivacaine that is hypobaric relative to CSF. This promotes cranial distribution of bupivacaine within the CSF and blockade of the higher spinal nerve roots, thus ensuring adequate extent of sensory block, even when administering doses as low as 10 mg of bupivacaine. This hypobaric bupivacaine solution is prepared by mixing 2 mL(milliliter) of isobaric 0.5% bupivacaine with 1 mL of sterile water. The investigators have demonstrated the efficacy of this for successful surgical anesthesia of adequate, but not excessive, duration in a recently concluded observational study. Notably, two subjects in the cohort of 60 patients received spinal anesthesia at the L5-S1 level. Both patients had adequate sensory block height and duration for commencement and completion of surgery without need for anesthetic supplementation. The investigator(s) have performed spinal anesthesia at the L5-S1 level in many other patients over the last 3 years with the same dose of hypobaric bupivacaine and have not encountered failure to date.

The purpose of this observational study is to determine the success rate of spinal anesthesia with low-dose (10 mg) hypobaric bupivacaine injected into the L5-S1 space in patients undergoing total hip or knee arthroplasty surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective unilateral total hip or knee arthroplasty under spinal anesthesia at TWH who are scheduled for inpatient overnight admission
* American Society of Anesthesiologists physical status class (ASA-PS) 1-3
* At least 20 years of age

Exclusion Criteria:

* Refusal to participate
* Inability to communicate due to language barrier or cognitive impairment
* Height > 200 cm
* Weight >120 kg
* Body mass index (BMI) >45 kg/m^2
* Contraindication or allergy to amide-type local anesthetic
* Contraindication to spinal anesthesia at the L5-S1 space (e.g., infection at the injection site, existing coagulopathy, severe spinal stenosis at higher vertebral levels)
* Previous spinal surgery in the lumbosacral spine
* Spinal anesthesia performed in the operating room rather than the block room
* Spinal anesthesia that includes administration of intrathecal opioids (e.g., morphine, fentanyl)
* Pre-existing sensory or motor impairment in the lower extremities
* Inability to identify the L5-S1 space with ultrasonography

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults aged at least 20 years having inpatient elective unilateral total hip or knee arthroplasty surgery
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2024-07-22 (Actual); Primary Completion 2025-03-20 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of successful spinal anesthesia | Assessed from time of spinal injection to surgery completion
  "Successful spinal anesthesia" is defined as the completion of surgery without conversion to general anesthesia, administration of supplemental opioids or surgical local anesthetic infiltration in the operating room to manage surgical pain.
Most cranial dermatomal level of sensory anesthesia achieved before surgery | Assessed every 5 minutes for the first 30 minutes after spinal injection
  A pinprick test using an 18G(gauge) blunt-tipped needle (BD Blunt Fill needle) will be performed on non-dependent and dependent sides to detect sensory loss over the torso and lower limbs. Sensation to pinprick testing in each dermatome will be categorized as normal ("sharp" sensation), analgesia ("dull" sensation), or anesthesia ("no" sensation).
  The most cephalad/cranial (upper) sensory block level of analgesia and anesthesia will be recorded based on the dermatomal map.
Time to reach the most cranial dermatomal level of sensory anesthesia before surgery | Assessed from time of spinal injection to surgery commencement
  The most cranial dermatomal level of sensory anesthesia will be determined based on the pinprick test.
Time to reach sensory anesthesia at level of T10 or higher before surgery, on the operative limb | Assessed from time of spinal injection to surgery commencement
  The dermatomal level of sensory anesthesia will be determined based on the pinprick test.
Time to reach sensory anesthesia at level of L1 or higher before surgery, on the operative limb | Assessed from time of spinal injection to surgery commencement
  The dermatomal level of sensory anesthesia will be determined based on the pinprick test.
Time to recovery of normal sensation at T10 or lower (also defined as duration of sensory analgesia at T10 or higher) in both lower limbs | Assessed at the end of surgery and every 30 minutes in the post-anesthesia care unit (PACU) or inpatient ward until a return of normal sensation in the T10 dermatome has been documented
  The dermatomal level of sensory anesthesia will be determined based on the pinprick test.
Time to normal sensation at L1 or lower (also defined as duration of sensory analgesia at L1 or higher) in both lower limbs | Assessed at the end of surgery and every 30 minutes in the PACU or inpatient ward until a return of normal sensation in the L2 dermatome has been documented on the day of surgery.
  The dermatomal level of sensory anesthesia will be determined based on the pinprick test.
Time to recovery of normal sensation at L2 or lower in both lower limbs | Assessed at the end of surgery and every 30 minutes in the PACU or inpatient ward until a return of normal sensation in the L2 dermatome has been documented on the day of surgery.
  The dermatomal level of sensory anesthesia will be determined based on the pinprick test.
Time to achieve complete motor block at hip, knee, ankle, and toes | Assessed every 5 minutes for the first 30 minutes after spinal injection
  The development of motor block will be assessed by assessing the ability to actively flex and extend at the hip, ankle, knee, and toes. This will be scored as either 1 (movement present and observed) or 0 (movement absent) at each joint on both lower extremities.
Time to regain ability to move hip, knee, ankle, and toes; and a score of 0 on the modified Bromage scale | Assessed at the end of surgery and every 30 minutes in the PACU or inpatient ward until full motor recovery has been achieved in both lower limbs on the day of surgery.
  Modified Bromage scale scores:
  0 - Able to move hip, knee, ankle and toes
  1. - Unable to move hip, able to move knee, ankle and toes
  2. - Unable to move hip and knee, able to move ankle and toes
  3. - Unable to move hip, knee and ankle, able to move toes
  4. - Unable to move hip, knee, ankle, or toes

SECONDARY OUTCOMES:
Time to scan, locate and mark the L5-S1 space | Assessed before surgery
  Time between first skin-probe contact to completion of skin markings.
Time to perform the spinal anesthetic | Assessed before surgery
  Time between injection of skin local anesthetic to completion of spinal anesthetic injection.
Number of needle passes | Assessed before surgery
  Each needle pass is defined as an insertion followed by a withdrawal of the spinal needle.
Incidence of adverse effects after spinal anesthesia | Assessed after the end of surgery and during the patient's stay in PACU or in-patient ward on the day of surgery.
  The following side-effects and adverse effects of spinal anesthesia will be assessed and recorded:
  i) Incidence of hypotension following spinal anesthesia and prior to intraoperative sedation
  ii) Incidence of postoperative nausea and vomiting (PONV) in the PACU, defined as need for administration of anti-emetic medication during the patient's stay in the PACU on the day of surgery.
  iii) Urinary retention (defined as need for urinary catheterization after surgery in PACU or in-patient ward on the day of surgery.
Patient satisfaction with anesthesia care, based on Likert scale | Assessed at the last study assessment visit, when regression to L2 has been documented either in PACU or in-patient ward on the day of surgery.
  Assessed using a 5-point Likert scale.
  1. Very dissatisfied
  2. Somewhat dissatisfied
  3. Neutral - neither satisfied nor dissatisfied
  4. Somewhat satisfied
  5. Very satisfied
  In the event of a score of 1-2 on the Likert scale, the patient will be asked to clarify the reasons for dissatisfaction with the anesthetic and how they think this could be improved with the following questions:
  i) "What did you not like about the anesthetic experience?" ii) "How could this be improved in the future?"
Patient satisfaction with anesthesia care, based on 3-response question | Assessed at the last study assessment visit, when regression to L2 has been documented either in PACU or in-patient ward on the day of surgery.
  Assessed using a 3-response question: "Would you choose to have the same anesthetic for similar surgery in the future?"
  Responses: Yes / Unsure / No
  In the event of a "No" response, the patient will be asked to clarify the reasons for dissatisfaction with the anesthetic and how they think this could be improved with the following questions:
  i) "What did you not like about the anesthetic experience?" ii) "How could this be improved in the future?"
Surgeon's perception of quality of intraoperative anesthesia | Assessed at the end of surgery and before the patient is transferred to PACU on the day of surgery.
  Surgeon's perception of the quality of anesthesia, in terms of the operating conditions provided by the spinal anesthetic. Assessed using a 3-point Likert scale:
  1. Poor (lowest score, worst outcome)
  2. Acceptable
  3. Good (highest score, best outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Ki Jinn Chin, MBBS,MMed,FRCPC, Principal Investigator — UHN
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No